CLINICAL TRIAL: NCT02041962
Title: Implementing Health Plan-Level Care Management for Solo & Small Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy M. Kilbourne, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R18HS021425-01A1 (AHRQ)
Record Dates: First submitted 2014-01-03; First posted 2014-01-22 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Bipolar Disorder; Depression
Keywords: Care Management; Chronic Care Model; Mood Disorders
MeSH Terms: conditions — Bipolar Disorder; Depression; Mood Disorders | interventions — Chronic Care Model

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Control (Active Comparator): Patients will receive their usual care from providers at their clinic. They will also receive in the mail a self-guided workbook.
  Interventions: Other: Educational Control
- Chronic Care Model for Mood Disorders (Experimental): Life Goals Collaborative Care
  Interventions: Behavioral: Chronic Care Model for Mood Disorders

INTERVENTIONS:
Behavioral: Chronic Care Model for Mood Disorders — The mood disorders CCM intervention ("Life Goals Collaborative Care") consists of: (a) a web-based patient self-management skills enhancement (CCM-1), (b) enhanced information flow and continuity of care via a care manager (CCM-2), and (c) decision support, or situation-specific evidence-based clinical practice guideline recommendations for providers (CCM-3). The CCM will be implemented utilizing telephonic contact with patients and providers by an Aetna care managers.The care managers will also use the Life Goals web portal as a guide for each session.
  Other Names: Life Goals Collaborative Care
  Arms: Chronic Care Model for Mood Disorders
Other: Educational Control
  Arms: Educational Control

SUMMARY:
This study will determine if a version of the chronic care model for individuals with mood disorders seen in small or solo practices can improve patient health.

DETAILED DESCRIPTION:
A 2010 HHS report highlighted the prevalence, morbidity, and cost associated with clusters of co-occurring chronic conditions, both physical and mental. The report also underscored the lack of sustainable treatment strategies for these afflicted individuals, and the difficulties in customizing patient-centered interventions.

Collaborative chronic care models (CCMs) are effective in treating chronic medical and mental illnesses at little to no net healthcare cost. To date CCMs have primarily been implemented at the facility level and primarily developed for and adopted by larger healthcare organizations. However, we have determined that the vast majority of primary care and behavioral health practices providing commercially insured care are far too small to implement such models. Health plan-level CCMs can address this unmet need.

Chronic mood disorders (e.g., bipolar disorders, depression) are common and are associated with extensive functional impairment, medical comorbidity, and personal and societal costs. While unipolar depression is more common, bipolar disorder is more costly on a per patient basis due to its chronic and severe nature. Moreover, bipolar disorder is the most expensive mental disorder for U.S. commercial health plans and employers. While evidence-based care parameters have been well established for mood disorders, quality of care and health outcomes in general mental health practice are suboptimal. The majority of these patients suffer from clusters of comorbid conditions, both physical and mental. Thus mood disorders represent optimal tracer conditions with which to improve management strategies for individuals with multiple chronic conditions.

Accordingly, we have partnered with Aetna Inc. to develop and implement a CCM designed to improve outcomes for persons with mood disorders for solo or small practices, with an eye towards developing a business case for a generalizable plan-level CCM for chronic disorders. We will conduct an RCT of a health plan-level CCM vs. education control. The population of interest will be Aetna beneficiaries across the country hospitalized for depression or bipolar disorder treated in solo or small primary care or behavioral health practices. Patients will be randomized to one year of outpatient treatment augmented by the CCM or education control, for a total of 344 participants. Practices participation in the study will be limited to completion of an organizational survey. We anticipate 172 practices to complete these surveys. CCM care management will be fully remote from practice venues and patients, implemented by existing providers (the Aetna care management center). A business case will be developed using the Replicating Effective Programs (REP) strategy that identifies generalizable facilitators for CCM spread and value added of CCMs to be vetted to key industry and policy stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Currently covered by Aetna's HMO or preferred provider products (for whom Aetna provides mental and medical inpatient, outpatient, and pharmacy benefits) for at least 6 months
* Recent (past 6-month) hospitalization for an acute psychiatric or partial hospital unit with a manic or depressive episode and confirmation of mood disorder diagnosis in the medical record (presence of one inpatient or two outpatient ICD-9 codes: 296.1x-296.8x in previous 6 months)
* Ability to speak and read English and provide informed consent
* Current principal outpatient prescribing provider is a solo practitioner or in a practice with <=3 providers.

Exclusion Criteria:

* No active substance intoxication
* No acute medical illness or dementia

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-07; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Kilbourne, PhD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Kilbourne AM, Prenovost KM, Liebrecht C, Eisenberg D, Kim HM, Un H, Bauer MS. Randomized Controlled Trial of a Collaborative Care Intervention for Mood Disorders by a National Commercial Health Plan. Psychiatr Serv. 2019 Mar 1;70(3):219-224. doi: 10.1176/appi.ps.201800336. Epub 2019 Jan 3. PMID 30602344
- [Derived] Kilbourne AM, Nord KM, Kyle J, Van Poppelen C, Goodrich DE, Kim HM, Eisenberg D, Un H, Bauer MS. Randomized controlled trial of a health plan-level mood disorders psychosocial intervention for solo or small practices. BMC Psychol. 2014 Nov 13;2(1):48. doi: 10.1186/s40359-014-0048-x. eCollection 2014. PMID 25520807

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 280 participants were consented and enrolled to participate. Of those 280 participants, only 238 completed the baseline survey and were randomized.
Groups:
- Educational Control: Patients will receive their usual care from providers at their clinic. They will also receive in the mail a self-guided workbook.
  Educational Control
Period: Overall Study
Arm/Group | Educational Control | Chronic Care Model for Mood Disorders
Started (Completed baseline and randomized) | 123 | 115
Participants Completing 6 mo. f/up | 69 | 44
Participants Completing 12 mo. f/up | 42 | 31
Completed | 42 | 31
Not Completed | 81 | 84
Not completed — Lost Aetna Coverage | 43 | 40
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 37 | 32
Not completed — Withdrawal by Subject | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Control | Chronic Care Model for Mood Disorders | Total
Number analyzed (Participants) | 123 | 115 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (13.2) | 42.8 (12.9) | 41.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 77 | 156
  Male | 44 | 38 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 94 | 99 | 193
  Not Available | 29 | 16 | 45
Region of Enrollment [Number; unit: participants]
  United States | 123 | 115 | 238
Health-related Quality of Life - Mental Health Component Score [Mean (Standard Deviation); unit: units on a scale] — Mental Health Quality of Life was measured using the 12-item Short Form Survey (SF-12). The SF-12 has a scale range of 0-100 with higher values representing better outcomes.
  units on a scale | 34.4 (15.2) | 36.9 (15.3) | 35.6 (15.2)
Mood Disorder Symptoms [Mean (Standard Deviation); unit: units on a scale] — Mood disorder symptoms were measured using the Patient Health Questionnaire (9-question). The PHQ-9 has a scale range of 0-27 with lower values representing better outcomes.
  units on a scale | 12.4 (6.1) | 13.0 (7.1) | 12.7 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life, as Measured by the Mental Health Component Score
Description: Mental Health Quality of Life was measured using the 12-item Short Form Survey (SF-12). The SF-12 has a scale range of 0-100 with higher values representing better outcomes.
Time Frame: 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Educational Control | Chronic Care Model for Mood Disorders
Number analyzed (Participants) | 42 | 31
score on a scale | 38.2 (9.6) | 43.2 (10.3)

2. Primary Outcome: Mood Disorder Symptoms, as Measured by the Patient Health Questionnaire (9-question)
Description: Mood disorder symptoms were measured using the Patient Health Questionnaire (9-question). The PHQ-9 has a scale range of 0-27 with lower values representing better outcomes.
Time Frame: 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Educational Control | Chronic Care Model for Mood Disorders
Number analyzed (Participants) | 42 | 31
score on a scale | 9.3 (4.2) | 7.6 (3.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 12-month period
Arm/Group | Educational Control | Chronic Care Model for Mood Disorders
All-Cause Mortality (participants affected / at risk) | 1/123 | 1/115
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/115
Other Adverse Events (participants affected / at risk) | 0/123 | 0/115

LIMITATIONS AND CAVEATS:
Dropout was substantial; the primary reason for subject dropout was disenrollment from Aetna coverage, as enrollment in Aetna was a study inclusion criterion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT02041962/Prot_SAP_000.pdf